CLINICAL TRIAL: NCT07300267
Title: A Phase 1, Randomized, Double-Blind, Active Comparator Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of a Novel Pneumococcal Vaccine in Children
Brief Title: A Clinical Study of Novel Pneumococcal Vaccine V118C in Children (V118C-002)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V118C-002
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- V118C (Stage 1) (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V118C administered at 12 to 15 months of age.
  Interventions: Biological: V118C (Stage 1)
- V118C (Stage 2) (Experimental): Participants will receive a single 0.5 mL IM injection of V118C administered at 2,4,6, and 12 months of age.
  Interventions: Biological: V118C (Stage 2)
- PCV20 (Stage 1) (Active Comparator): Participants will receive a single 0.5 mL IM injection of PCV20 administered at 12 to 15 months of age.
  Interventions: Biological: PCV20 (Stage 1)
- PCV20 (Stage 2) (Active Comparator): Participants will receive a single 0.5 mL IM injection of PCV20 administered at 2,4,6, and 12 months of age.
  Interventions: Biological: PCV20 (Stage 2)

INTERVENTIONS:
Biological: V118C (Stage 1) — IM administration of V118C
  Arms: V118C (Stage 1)
Biological: V118C (Stage 2) — IM administration of V118C
  Arms: V118C (Stage 2)
Biological: PCV20 (Stage 1) — IM administration of PCV20
  Arms: PCV20 (Stage 1)
Biological: PCV20 (Stage 2) — IM administration of PCV20
  Arms: PCV20 (Stage 2)

SUMMARY:
Researchers are looking for new vaccines to prevent pneumococcal disease, which is any infection in the lungs or other parts of the body that is caused by a type of bacteria called Streptococcus pneumoniae. V118C is a new vaccine designed to help prevent disease from Streptococcus pneumoniae bacteria.

This study will look at V118C in toddlers and infants. The goal of the study is to learn how safe V118C is for children and how well they tolerate it.

DETAILED DESCRIPTION:
Stage 1 of the study will be conducted in toddlers enrolled at 12 through 15 months of age who previously completed a primary 3-dose infant series with a licensed pneumococcal conjugate vaccine (PCV). Stage 2 will be conducted in infants enrolled at approximately 2 months of age, who will receive the 3+1 schedule (3 infant doses followed by a toddler dose).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

Stage 1:

* Is previously vaccinated with 3 routine infant doses of Pneumococcal 20-valent conjugate vaccine (PCV20)
* Is 12 through 15 months of age

Stage 2:

- Is approximately 2 months of age

Both Stages:

* Was born at full term (gestational age greater than or equal to 37 weeks)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

Stage 1:

- Has received a PCV dose at 10 months of age and older

Stage 2:

* Has received prior administration of any pneumococcal vaccine

Both stages:

* Has a history of invasive pneumococcal disease (IPD)
* Has a known hypersensitivity to any component of V118C or PCV20 including diphtheria toxoid

Ages: 2 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2028-10-24 (Estimated); Study Completion 2029-05-25 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Percentage of Participants With Immediate Adverse Events (AEs) Following Vaccination | Up to approximately 30 minutes postvaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants with immediate AEs following vaccination will be reported.
Stage 1: Percentage of Participants With Solicited Injection-Site Adverse Events (AEs) | Up to approximately 7 days postvaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A solicited AE is a predefined event that participants legally acceptable representative (LAR) are specifically asked about and record on their electronic vaccine report card (eVRC). Solicited injection-site AEs include redness, swelling, pain or tenderness and hard lump. Percentage of participants with solicited injection-site AEs will be reported.
Stage 1: Percentage of Participants With Solicited Systemic AEs | Up to approximately 7 days postvaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A solicited AE is a predefined event that participants LAR are specifically asked about and record on their eVRC. Solicited systemic AEs include irritability, drowsiness, appetite lost, hives or welts, and fever. Percentage of participants with solicited systemic AEs will be reported.
Stage 1: Percentage of Participants With Unsolicited Systemic or Injection-Site AEs | Up to approximately 28 days postvaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE is an event that is not solicited using a eVRC and that is communicated by a participant. Percentage of participants with unsolicited Systemic or Injection-Site AEs will be reported.
Stage 1: Percentage of Participants With Serious Adverse Events (SAEs) | Up to approximately 12 months postvaccination
  A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Percentage of participants with one or more SAEs will be reported.
Stage 1: Percentage of Participants With Medically Attended AEs (MAAEs) | Up to approximately 12 months postvaccination
  A MAAE is defined as an adverse event in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency department visit, office visit, or an urgent care visit with any medical personnel for any reason. Percentage of participants with MAAEs will be reported.
Stage 2: Percentage of Participants With Immediate AEs Following Vaccination | Up to approximately 30 minutes after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants with immediate AEs following vaccination will be reported.
Stage 2: Percentage of Participants With Solicited Injection-Site AEs | Up to approximately 7 days after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A solicited AE is a predefined event that participants LAR are specifically asked about and record on their eVRC. Solicited injection-site AEs include redness, swelling, pain or tenderness and hard lump. Percentage of participants with solicited injection-site AEs will be reported.
Stage 2: Percentage of Participants With Solicited Systemic AEs | Up to approximately 7 days after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A solicited AE is a predefined event that participants LAR are specifically asked about and record on their eVRC. Solicited systemic AEs include irritability, drowsiness, appetite lost, hives or welts, and fever. Percentage of participants with solicited systemic AEs will be recorded.
Stage 2: Percentage of Participants With Unsolicited Systemic or Injection-Site AEs | Up to approximately 28 days after each vaccination
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An unsolicited AE is an event that is not solicited using a eVRC and that is communicated by a participant. Percentage of participants with unsolicited Systemic or Injection-Site AEs will be reported.
Stage 2: Percentage of Participants With SAEs | Up to approximately 12 months postdose 4
  A SAE is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Percentage of participants with one or more SAEs will be reported.
Stage 2: Percentage of Participants With MAAEs | Up to approximately 12 months postdose 4
  A MAAE is defined as an adverse event in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency department visit, office visit, or an urgent care visit with any medical personnel for any reason. Percentage of participants with MAAEs will be reported.

SECONDARY OUTCOMES:
Stage 1: Geometric Mean Concentrations (GMCs) of Serotype-Specific Immunoglobulin G (IgG) | Up to approximately 30 days post vaccination
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay. GMCs of Serotype-specific IgG at 30 days postvaccination with V118C and PCV20 will be reported.
Stage 1: Ratio of GMCs of Serotype-Specific IgG of V118C to PCV20 [V118C/PCV20] | Approximately Day 30 postvaccination
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay. Ratio of GMCs of serotype-specific IgG of V118C to PCV20 will be reported.
Stage 1: Geometric Mean Fold Rises (GMFRs) of Serotype-Specific Immunoglobulin G (IgG) | Day 1 (Baseline) and approximately Day 30 postvaccination
  Geometric mean fold rise (GMFR) is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline. GMFRs of serotype-specific IgG from baseline (Day 1) to Day 30 with V118C and PCV20 for IgG responses will be reported.
Stage 1: Percentage of Participants With a ≥ 4-fold Rise for Serotype Specific IgG Concentrations | Day 1 (Baseline) and approximately Day 30 postvaccination
  The percentage of participants with ≥4-fold rise from baseline (Day 1) to Day 30 with V118C and PCV20 for IgG responses will be reported.
Stage 2: Percentage of Participants With IgG ≥0.35 μg/mL (Response Rates) for Serotype Specific IgG Concentrations at 30 Days Postdose 3 | Up to approximately 30 days postdose 3
  Percentage of participants with IgG ≥0.35 μg/mL (response rates) for each serotype at 30 days postdose 3 (PD3) with V118C and PCV20 will be reported will be reported.
Stage 2: Percentage of Participants With IgG ≥0.35 μg/mL (Response Rates) for Serotype Specific IgG Concentrations at 30 Days Predose 4 | Up to approximately 6 months post dose 3
  Percentage of participants with IgG ≥0.35 μg/mL (response rates) for each serotype at predose 4 (PD4) with V118C and PCV20 will be reported.
Stage 2: Percentage of Participants With IgG ≥0.35 μg/mL (Response Rates) for Serotype Specific IgG Concentrations at 30 Days Postdose 4 | Up to approximately 30 days postdose 4
  Percentage of participants with IgG ≥0.35 μg/mL (response rates) for each serotype at 30 days postdose 4 with V118C and PCV20 will be reported.
Stage 2: Difference in the Response Rates [V118C minus PCV20] for Each Serotype at 30 Days Postdose 3 | Up to approximately 30 days postdose 3
  Difference in the response rates [V118C minus PCV20] for each serotype at 30 days postdose 3 with V118C and PCV20 will be reported.
Stage 2: Difference in the Response Rates [V118C Minus PCV20] for Each Serotype at 30 Days Postdose 4 | Up to approximately 30 days postdose 4
  Difference in the response rates [V118C minus PCV20] for each serotype at 30 days postdose 4 with V118C and PCV20 will be reported.
Stage 2: GMCs of Serotype-Specific IgG at 30 Days Postdose 3 | Up to approximately 30 days postdose 3
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay. GMCs of serotype-specific IgG at 30 days postdose 3 with V118C and PCV20 will be reported.
Stage 2: GMCs of Serotype-Specific IgG at 30 Days Predose 4 | Up to approximately 6 months post dose 3
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay. Serotype-specific IgG GMCs at 30 days predose 4 with V118C and PCV20 will be reported.
Stage 2: GMCs of Serotype-Specific IgG at 30 Days Postdose 4 | Up to approximately 30 days postdose 4
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay. Serotype-specific IgG GMCs at 30 days postdose 4 with V118C and PCV20 will be reported.
Stage 2: Ratio of Serotype-Specific IgG GMCs of V118C to PCV20 [V118C/PCV20] at 30 Days Postdose 3 | Up to approximately 30 days postdose 3
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay. Ratio of serotype-specific IgG GMCs of V118C to PCV20 [V118C/PCV20] at 30 days postdose 3 will be reported.
Stage 2: Ratio of Serotype-Specific IgG GMCs of V118C to PCV20 [V118C/PCV20] at 30 Days Postdose 4 | Up to approximately 30 days postdose 4
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (Pn ECL) assay. Ratio of serotype-specific IgG GMCs of V118C to PCV20 [V118C/PCV20] at 30 days postdose 4 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- United States (8):
  - Madera Family Medical Group ( Site 1004), Madera, California
  - Cotton O'Neil Research Center ( Site 1039), Topeka, Kansas
  - University of Louisville, Norton Children's Research Institute ( Site 1005), Louisville, Kentucky
  - Tribe Clinical Research, LLC-Pediatrics ( Site 1008), Greenville, South Carolina
  - Tribe Clinical Research, LLC-Pediatrics ( Site 1001), Spartanburg, South Carolina
  - Epic Medical Research - Carrollton ( Site 1038), Carrollton, Texas
  - University of Texas Medical Branch ( Site 1020), League City, Texas
  - Pediatric Research of Charlottesville, LLC ( Site 1012), Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com